CLINICAL TRIAL: NCT04247984
Title: An Efficacy and Safety Study of mXELIRI Versus. FOLFIRI + Bevacizumab Therapy as First-line Chemotherapy in Metastatic Colorectal Cancer
Brief Title: A Comparison of mXELIRI Regimen and FOLFIRI Combined Bevacizumab Regimen as First-line Chemotherapy Regimen for Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences (Other)
Collaborators: Beijing Hospital (Other Government); Henan Cancer Hospital (Other Government); Liaoning Cancer Hospital & Institute (Other); Jiangsu Cancer Institute & Hospital (Other)
Responsible Party: Principal Investigator, Aiping Zhou, Chief physician, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCC-000583
Record Dates: First submitted 2020-01-23; First posted 2020-01-30 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Metastatic Colorectal Cancer
Keywords: XELIRI; FOLFIRI
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab; Capecitabine; Irinotecan; Fluorouracil

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mXELIRI+ Bevacizumab (Experimental)
  Interventions: Biological: Bevacizumab; Drug: Capecitabine; Drug: Irinotecan
- FOLFIRI + Bevacizumab (Active Comparator)
  Interventions: Biological: Bevacizumab; Drug: Irinotecan; Drug: 5-FU; Drug: CF

INTERVENTIONS:
Biological: Bevacizumab — 5 mg/kg intravenously administered on day 1 of a 2-week cycle.
  Other Names: Avastin
Drug: Capecitabine — 2000mg/m2/day oral on day 1 to day 10 of a 2-week cycle.
  Other Names: Xeloda
  Arms: mXELIRI+ Bevacizumab
Drug: Irinotecan — 180 mg/m2 intravenously administered on day 1 of a 2-week cycle.
  Other Names: CPT-11
  Arms: FOLFIRI + Bevacizumab
Drug: 5-FU — 400 mg/m2 intravenous bolus on day 1 and 2400 mg/m2 continuous infusion over 44 hours of a 2-week cycle.
  Other Names: Fluorouracil
  Arms: FOLFIRI + Bevacizumab
Drug: CF — 300 mg/m2 intravenously administered on day 1 of a 2-week cycle.
  Arms: FOLFIRI + Bevacizumab
Drug: Irinotecan — 150 mg/m2 intravenously administered on day 1 of a 2-week cycle.
  Other Names: CPT-11
  Arms: mXELIRI+ Bevacizumab

SUMMARY:
This is a Phase II, multicenter，randomized, two arms, open-labeled, controlled clinical trial. This trial was conducted to evaluate the efficacy and safety of bevacizumab (Avastin®) plus mXELIRI compared with bevacizumab (Avastin®) plus FOLFIRI as first-line treatment in patients with metastatic colorectal cancer (mCRC).

DETAILED DESCRIPTION:
This is a Phase II, multicenter，randomized, two arms, open-labeled, controlled clinical trial. This trial was conducted to evaluate the efficacy and safety of bevacizumab (Avastin®) plus mXELIRI compared with bevacizumab (Avastin®) plus FOLFIRI in not previously treated patients with metastatic colorectal cancer (mCRC). In experimental group, untreated patients with metastatic colorectal cancer will receive Irinotecan 150 mg/m2 (D1, q2w) , Xeloda 2000mg/m2 (D1-10, q2w) and bevacizumab 5mg/kg (D1, q2w) for 6-9 cycles as the first-line treatment. While in control group, patients with metastatic colorectal cancer will receive Irinotecan 180 mg/m2 (D1, q2w) , CF 300mg/m2 (D1 q2w), 5FU 400mg/m2, D1 2400 mg/m2, civgtt 44h (q2w) and bevacizumab 5mg/kg (D1, q2w) for 6-9 cycles as the first-line treatment.The primary endpoint is progression-free survival. Overall survival, Objective Response rate, adverse event and life quality will be assessed as secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent;
2. ECOG≤1;
3. Age≥18；
4. Histologically or cytologically confirmed unresectable metastatic colorectal cancer with no previous chemotherapy or molecular targeted therapy;
5. At least one evaluable lesion per RECIST (Response Evaluation Criteria in Solid Tumors) 1.1;
6. life expectancy >12 weeks;
7. Adequate bone marrow and organ function. Hb≥9 G/L; Absolute neutrophil ≥ 1.5 G/L; PLT ≥100 G/L ;ALT/AST ≤2 ULN or ≤5ULN with liver metastases;ALP ≤2.5 ULN or ≤5ULN with liver metastases or ≤10ULN with bone metastases ; TBIL ≤1.5 ULN; Cr≤1.0 ULN;
8. Urinary protein excretion < 2+ (dipstick). If > or equal 2+ proteinuria is detected with dipstick, a 24-hour period urine test will be performed and the result should be < or equal to 1 g/24 hours to permit the inclusion of the patient in the clinical trial.

Exclusion Criteria:

1. Pregnant or lactating women；
2. Sexually active women (of childbearing potential) or men unwilling to adopt an effective method of birth control during the course of the study；
3. Previous treatment with Irinotecan or anti-VEGF antibodies;
4. Any previous malignancy within 5 years prior to study entry, except for cured basal cell carcinoma of skin or carcinoma-in-situ of the uterine cervix;
5. History of acute coronary syndromes (including myocardial infarction and unstable angina) within 6 months prior to study entry, or history or evidence of current ≥ Class II congestive heart failure as defined by New York Heart Association (NYHA);
6. Uncontrolled hypertension and severe arrhythmia requiring drug treatment;
7. Present with non-healing fractures or wounds of skin;
8. History of previous abdominal fistula, gastrointestinal perforation or intra-abdominal abscesses within 6 months before randomization;
9. Major surgery, open surgical biopsy or significant traumatic injury within 4 weeks or needle biopsy within 7 days before randomization before randomization；
10. Evidence or history of bleeding diathesis or coagulopathy；
11. Known or suspected allergy or hypersensitivity to any component of Bevacizumab, xeloda, irinotecan, or 5-FU/LV;
12. Clinical or radiological evidence of CNS metastases;
13. History of unexpected serious adverse events to fluoropyrimidine treatments or known dihidropyrimidine dehydrogenase (DPD) deficiency;
14. Patients subjected to organ allografts who require immunosuppressive treatment;
15. Prior adjuvant or neoadjuvant treatment for metastatic colorectal cancer is allowed, as long as it has concluded at least 6 months before beginning the treatment of the study;
16. If adjuvant treatment has previously been administered, the patients cannot have shown progression of the disease during treatment nor during the 6 months following termination thereof;
17. Prior radiotherapy is allowed if it has not been administered in the target lesions selected for this study, unless progression of said lesions in the irradiated field is documented, and as long as treatment has concluded at least 4 weeks before beginning the study;
18. Prior surgical treatment of the disease in stage IV is allowed;
19. Use of full dose of oral or parenteral anticoagulants ( at least 10 days before the initial study treatment or thrombolytic agents. Low dose of warfarin is allowed, with an INR ≤ 1.5;
20. Subject requiring chronic use of high dose aspirin (> 325 m/day) or non-steroidal anti-inflammatory treatment ;
21. Received any investigational drug or agent/ procedure, i.e. participation in another treatment trial within 4 weeks of randomisation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 6 Months
  Time from the date of enrollment to the earlier of the date of confirmed progression or death from any cause.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | 6 Months
  Proportion of eligible patients with measurable lesions with a best overall response of CR or PR assessed by the attending physician.
Overall survival (OS) | 1 Year
  Time from the date of enrollment to death from any cause.
Incidence of Adverse Events | 6 Months
  The incidence of adverse events as graded by NCI-CTCAE v 4.0.
Quality of life (QoL) Questionnaire | 6 Months
  Determined by European Organization for Research and Treatment of Cancer (EORTC) Quality-of-Life Questionnaire-Core 30 (QLQ-C30) Score

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital & Institute, Chinese Academy of Medical Sciences, Beijing, China